CLINICAL TRIAL: NCT00331240
Title: 24-Hour Intraocular Pressure (IOP) Control With Travoprost/Timolol Fixed Combination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A1457
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Primary Open Angle Glaucoma; Exfoliation Syndrome
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome | interventions — Travoprost; Lubricant Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: travoprost/timolol fixed combination
Drug: placebo (artificial tears)

SUMMARY:
The purpose of this study is to compare the short-term (8 week) mean 24-hour intraocular pressure control and safety of TravTim fixed combination given once in the evening with placebo once in the morning versus TravTim given once in the morning with placebo once in the evening in patients with open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* POAG
* Exfoliation syndrome

Exclusion Criteria:

* Advanced glaucoma

Ages: 29 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2006-03; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AGP Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, A University Dept of Ophthalmology, AHEPA Hospital
Locations (1):
- Glaucoma Unit, A University Dept of Ophthalmology, AHEPA Hospital, Thessaloniki, Greece